CLINICAL TRIAL: NCT05618795
Title: " Comparative Evaluation of Aggressive Gap Arthroplasty With Minimal Gap Arthroplasty in the Management of TMJ Ankylosis "
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PGIDS/BHRC/22/41 NILESH BAGDE
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Arthoplasty
Keywords: Gap Arthoplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aggresive gap arthoplasty (Other): control group- aggressive gap arthroplasty(15 to 20 mm) for management of TMJ ankyosis
  Interventions: Other: minimal gap arthoplasty v/s aggressive gap arthoplasty
- minimal gap arthoplasty (Active Comparator): experimental group-minimal gap arthroplasty(5 to 8mm) for management of TMJ ankylosis
  Interventions: Other: minimal gap arthoplasty v/s aggressive gap arthoplasty

INTERVENTIONS:
Other: minimal gap arthoplasty v/s aggressive gap arthoplasty — Comparative evaluation of aggressive gap arthroplasty with minimal gap arthroplasty in the management of TMJ ankylosis

SUMMARY:
the most commonly used protocol in the management of TMJ ankylosis is Kabans protocol in which 1.5 to 2 cm aggressive resection of bone is recommended which may lead to gap between cranial base and condyle of mandible.1 However, there are certain disadvantages associated with aggressive gap arthroplasty such as pseudo articulation with shortening of the mandibular ramus, premature occlusion on the affected side with a contralateral open bite in unilateral cases,2 in bilateral cases gagging of the posterior teeth and anterior open bite.3 Few studies in the literature available agreed that minimum gap arthroplasty i.e. 5 to 8 mm of gap is sufficient for TMJ movements in all planes and recurrence of ankylosis is likely to be prevented by interposed material (graft)4 .So, a randomized control study to compare outcomes of minimal gap arthroplasty with aggressive gap arthroplasty for management of TMJ ankylosis is planned.

DETAILED DESCRIPTION:
A standardize protocol for each patient will be followed that comprises of case selection, clinincal evaluation, radiographic assessment,treatment planning and measurement of varius parameters.

* Medical and Dental history of the patient will be obtained.
* A written consent form signed by the patient, will be obtained.
* Case evaluation will be done which will include clinical and radiographic evaluation Based on the case evaluation, surgical treatment of ankylosis will be performed . patient will be randomized into the following two groups. Group A -minimal gap arthroplasty for management of Tmj ankylosis Group B -aggressive gap arthroplasty for management of TMJ ankylosis A minimum of 6 subjects per group completing the study would be giving a good external validity to the present study.

  1. All the patients were evaluated with history, clinical and radiological examinations (panoramic and CT scans). Informed consent will be obtaine from all the patients.
  2. In both groups, all the patients will be operated by an experienced surgeon.The data acquisition will be done by a resident who will be kept blind for group allocation.

  3. In group 1 cases treatment of TMJ ankylosis will be done by minimal gap arthroplasty and in group 2 cases treatment of TMJ ankylosis will be done by aggressive gap arthroplasty 4. both groups cases will be evaluated preoperatively ,intraoperatively and postoperatively Follow-up visits will be at 1, 3, and 6 months 5. preoperative and postoperative evaluation will be done clinically ( mouth opening ,protrusive movement, laterotrusive movement ) , radiologically (OPG, CTscan) .

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy adult(ASA Classification I-II)
* Any age group
* Sawhneys classification type IV
* Unilateral ankylosis
* Written informed consent

Exclusion Criteria:

* Any syndromic patient
* Recurrence cases
* Sawhneys classification type I,II,III

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
mouth opening | T0- preoperatively
  maximal interincisal distance on opening mouth widely.
mouth opening | T1- 24hr after surgical intervention
  maximal interincisal distance on opening mouth widely.
mouth opening | T2- 1 month after surgical intervention
  maximal interincisal distance on opening mouth widely.
mouth opening | T3- 3 month after surgical intervention
  maximal interincisal distance on opening mouth widely.
mouth opening | T4- 6 month after surgical intervention
  maximal interincisal distance on opening mouth widely.

SECONDARY OUTCOMES:
Protrusive movement | T0- preoperatively
  maximal protrusive movement on mandibular advancement
Protrusive movement | T1- 24hr after surgical intervention
  maximal protrusive movement on mandibular advancement
Protrusive movement | T2- 1 month after surgical intervention
  maximal protrusive movement on mandibular advancement
Protrusive movement | T3- 3 month after surgical intervention
  maximal protrusive movement on mandibular advancement
Protrusive movement | T4- 6 month after surgical intervention
  maximal protrusive movement on mandibular advancement
Laterotrusive movement | T0- preoperatively
  maximal lateral movement on mandibular excursion
Laterotrusive movement | T1- 24hr after surgical intervention
  maximal lateral movement on mandibular excursion
Laterotrusive movement | T2- 1 month after surgical intervention
  maximal lateral movement on mandibular excursion
Laterotrusive movement | T3- 3 month after surgical intervention
  maximal lateral movement on mandibular excursion
Laterotrusive movement | T4- 6 month after surgical intervention
  maximal lateral movement on mandibular excursion
Any complication | T0- preoperatively
  Any complication after surgery
Any complication | T1- 24hr after surgical intervention
  Any complication after surgery
Any complication | T2- 1 month after surgical intervention
  Any complication after surgery
Any complication | T3- 3 month after surgical intervention
  Any complication after surgery
Any complication | T4- 6 month after surgical intervention
  Any complication after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Pgids, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No